CLINICAL TRIAL: NCT05672719
Title: Hemodynamic Testing Strategies to Assess Pulmonary Hypertension and Right Ventricular Function in Heart Failure Patients
Brief Title: Hemodynamic Testing Strategies to Assess Pulmonary Hypertension in Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor
Other Study IDs: G21-0031553
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Right Heart Catheterization — Procedure

SUMMARY:
The goal of this observational study is to learn about heart function and high lung blood pressure in patients with heart failure. The main question[s] it aims to answer are whether we can improve the ability to predict patients who will have complications after they receive treatment including heart transplant and left ventricular assist devices.

DETAILED DESCRIPTION:
Prospective cohort study of patients with heart failure with reduced ejection fraction that are referred for diagnostic right heart catheterization as part of their evaluation for candidacy for advanced heart failure therapies.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 years or older
* Heart failure with reduced ejection fraction (<40%)
* referred for RHC at our centre for evaluation of candidacy for advanced HF therapies.

Exclusion Criteria:

Severe valvular or complex congenital heart disease Short-term mechanical circulatory support for progressive cardiogenic shock (e.g. extracorporeal membrane oxygenation) Acute coronary syndrome or revascularization occurred within 7 days prior to the RHC.

Pregnant or breast-feeding Known hypersensitivity to sodium nitroprusside Advanced liver dysfunction Reduced capacity or inability to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients assessed in the advanced heart failure program for heart transplant candidacy at the University of Toronto referred for right heart catheterization.
Sampling Method: Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Mean pulmonary artery pressure | First study 1 day visit
  Hemodynamic measurement
right ventricular end systolic elastance | First study 1 day visit
  Hemodynamic measurement
pulmonary arterial elastance | First study 1 day visit
  hemodynamic measurement

SECONDARY OUTCOMES:
Right ventricular failure after heart transplant | 1 year
  Clinical outcome
Right ventricular failure after left ventricular assist device | 1 year
  Clinical outcome

OTHER OUTCOMES:
right ventricular pulmonary arterial elastance coupling response to vasodilator | First study 1 day visit
  Hemodynamic measurement

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Mak, MD PhD, Principal Investigator — University of Toronto
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Agreements to share participant data can be requested after study completion and publication.